CLINICAL TRIAL: NCT07094451
Title: Virtual Reality for Pain Control During US-guided Needle Procedures in Obstetric Patients: A Prospective Pilot Study
Brief Title: Virtual Reality for Pain Control in US-Guided Obstetric Needle Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Professor and Vice Chair of Education for the Department of Anesthesiology, Pain, & Perioperative Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-25-00020
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Procedural Pain
Keywords: Virtual reality; Procedural anxiety; Ultrasound-guided; Obstetric patients; Non-pharmacologic pain control; Immersive distraction
MeSH Terms: conditions — Pain, Procedural | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without Virtual Reality (VR) (Active Comparator): Standard of care procedure without virtual reality.
  Interventions: Procedure: Ultrasound
- Patients with Virtual Reality (Experimental): Ultrasound-guided (US-Guided) procedure with virtual reality.
  Participants will wear a Meta Quest 2 virtual reality headset during their ultrasound-guided needle procedure.
  Interventions: Device: Virtual Reality; Procedure: Ultrasound

INTERVENTIONS:
Device: Virtual Reality — Meta Quest 2 virtual reality headset. The VR experience includes an interactive, immersive environment with classical music and wrist-controlled movement to match floating visual cues to a beat. The experience is designed to be soothing and require minimal movement.
  Arms: Patients with Virtual Reality
Procedure: Ultrasound — Ultrasound-guided (US-Guided) procedure

SUMMARY:
This is a single-site randomized controlled pilot study at Mount Sinai Hospital evaluating the effect of virtual reality on procedural pain and anxiety in obstetric patients undergoing ultrasound-guided needle procedures. Patients will be randomized to receive either VR or standard care during the procedure and complete validated questionnaires assessing pain, anxiety, intervention acceptability, and satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18
* English-speaking
* Undergoing ultrasound-guided needle procedure at Mount Sinai

Exclusion criteria:

* History of seizures
* Severe motion sickness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Short-form McGill Pain Questionnaire | Immediately post-procedure
  The Short-form McGill Pain Questionnaire (SF-MPQ) is used to assess procedural pain and its qualities, such as 'sharpness.' The total score ranges from 0 to 45, with higher scores indicating more pain. It includes subscales for Sensory (0-33), Affective (0-12), a Visual Analogue Scale (0-10), and Present Pain Intensity (0-5).

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Immediately post-procedure (procedure lasts approximately 20 minutes)
  This is a short, 4-question survey that helps the research team understand how acceptable participants found the use of virtual reality (VR) during their procedure. Participants rate each statement (ex: "The VR intervention meets my approval") on a scale from 1 (completely disagree) to 5 (completely agree). The total score ranges from 4 to 20, with higher scores indicating greater acceptability of the VR experience.
State-Trait Anxiety Inventory (STAI) | Immediately Pre-procedure and immediately post-procedure (procedure lasts approximately 20 minutes)
  The STAI is a 20-item instrument assessing anxiety before and after procedure. Each item is rated on a 4-point scale from 1-4.
  Total scale range from 20 to 80, with higher scores indicating higher state anxiety.
Visual Analog Scale for Satisfaction | Immediately post-procedure (procedure lasts approximately 20 minutes)
  This is a simple one-question survey where participants rate how satisfied they were with their overall procedure experience. They will mark their satisfaction on a scale from 1 to 10, where 1 means "not satisfied at all" and 10 means "completely satisfied." The total score ranges from 1 to 10, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Obstetrics and Gynecology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a single-site, small-scale pilot study that does not include the collection of biospecimens or long-term follow-up data. The data collected are limited to de-identified questionnaire responses.